CLINICAL TRIAL: NCT01457924
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-Group, Dose-Ranging Study to Investigate the MRI Efficacy and Safety of Six Months' Administration of Ofatumumab in Subjects With Relapsing-Remitting Multiple Sclerosis (RRMS)
Brief Title: Ofatumumab Subcutaneous Administration in Subjects With Relapsing-Remitting Multiple Sclerosis
Acronym: MIRROR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112831
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis; Ofatumumab
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — ofatumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort 1 (Experimental): Placebo and one dose of Ofatumumab 3mg over 24 weeks
  Interventions: Drug: Ofatumumab 3mg; Drug: Placebo
- Cohort 2 (Experimental): Two doses of Ofatumumab 3mg over 24 weeks
  Interventions: Drug: Ofatumumab 3mg; Drug: Placebo
- Cohort 3.1 (Experimental): Two doses of Ofatumumab 30mg over 24 weeks
  Interventions: Drug: Ofatumumab 30mg; Drug: Placebo
- Cohort 3.2 (Experimental): Conditioning dose of Ofatumumab 3mg at randomization, two doses of Ofatumumab 30mg over 24 weeks
  Interventions: Drug: Ofatumumab 3mg; Drug: Ofatumumab 30mg; Drug: Placebo
- Cohort 4.1 (Experimental): Two doses of Ofatumumab 60mg over 24 weeks
  Interventions: Drug: Ofatumumab 60mg; Drug: Placebo
- Cohort 4.2 (Experimental): Conditioning dose of Ofatumumab 3mg at randomization, two doses of Ofatumumab 60mg over 24 weeks
  Interventions: Drug: Ofatumumab 3mg; Drug: Ofatumumab 60mg; Drug: Placebo
- Cohort 5.1 (Experimental): Six doses of Ofatumumab 60mg over 24 weeks
  Interventions: Drug: Ofatumumab 60mg; Drug: Placebo
- Cohort 5.2 (Experimental): Conditioning dose of Ofatumumab 3mg at randomization, six doses of Ofatumumab 60mg over 24 weeks
  Interventions: Drug: Ofatumumab 3mg; Drug: Ofatumumab 60mg

INTERVENTIONS:
Drug: Ofatumumab 3mg — 3mg of investigational product
  Arms: Cohort 1; Cohort 2; Cohort 3.2; Cohort 4.2; Cohort 5.2
Drug: Ofatumumab 30mg — 30mg of investigational product
  Arms: Cohort 3.1; Cohort 3.2
Drug: Ofatumumab 60mg — 60mg of investigational product
  Arms: Cohort 4.1; Cohort 4.2; Cohort 5.1; Cohort 5.2
Drug: Placebo — Placebo
  Arms: Cohort 1; Cohort 2; Cohort 3.1; Cohort 3.2; Cohort 4.1; Cohort 4.2; Cohort 5.1

SUMMARY:
Ofatumumab is a novel Immunoglobulin 1ĸ ( IgG1ĸ) lytic monoclonal antibody (mAb) that specifically binds to the human Cluster of Differentiation 20 (CD20) antigen of which expression is restricted to B lymphocytes from the pre-B cell stage to the plasmacytoid immunoblast stage only. A recent trial with an anti-CD20 mAb (rituximab) demonstrated that targeting B-cells reduces the number of gadolinium-enhancing (GdE) T1 lesions and the relapse rate in relapsing-remitting multiple sclerosis (RRMS). Ofatumumab has been shown to be both well tolerated and efficacious in several indications, including a small, placebo-controlled trial in RRMS using an intravenous (IV) formulation.

This double-blind, placebo-controlled, parallel-group study will investigate the safety and efficacy of a subcutaneous formulation of ofatumumab in the treatment of subjects with RRMS. The primary objective of the study is to investigate the efficacy as assessed by magnetic resonance imaging. Other objectives will include evaluation of tolerability/safety, dose-response relationship, pharmacokinetics, pharmacodynamics, exposure-response, as well as other clinical endpoints.

DETAILED DESCRIPTION:
Ofatumumab is a novel immunoglobulin G (IgG) 1ĸ lytic monoclonal antibody (mAb) that specifically binds to the human CD20 antigen of which expression is restricted to B lymphocytes from the pre-B cell stage to the plasmacytoid immunoblast stage only. A recent trial with rituximab demonstrated that targeting B-cells reduces the number of gadolinium-enhancing (GdE) T1 lesions and the relapse rate in Relapsing-Remitting Multiple Sclerosis (RRMS). The intravenous (IV) formulation of ofatumumab has been shown to be both well-tolerated and efficacious in Phase I/II & III clinical trials within in B-cell Chronic Lymphocytic Leukemia (B-CLL), non-Hodgkin's Follicular Lymphoma (FL), and active Rheumatoid Arthritis (RA). A Phase II study of ofatumumab in Relapsing Remitting Multiple Sclerosis (RRMS) subjects, OMS115102 (also known as Study GEN414) is ongoing as of the development of this protocol. The primary objective of the OMS115102 protocol was to investigate the safety of a range of doses (100mg, 300 mg, and 700 mg) of ofatumumab in RRMS subjects, using an IV formulation. The treatment period for OMS115102 has been completed; there are currently 4 subjects ongoing in the Individualized Follow up Phase. In the Week 0 to 24 period the majority of subject who were exposed to active treatment with ofatumumab (active/placebo) had Cluster of Differentiation 19 (CD19+) and CD20+ levels that were suppressed to zero; recovery started for the 100 mg and 300 mg active/placebo groups, at approximately, 12 and 20 weeks after discontinuation of dosing with ofatumumab, respectively. In the 700 mg active/placebo group, all but one subject had a persistent and complete CD19+ suppression at Week 24. In the Week 24 to 48 period, when those who had previously been exposed to placebo were treated with ofatumumab (placebo/active), the majority of the subjects treated with ofatumumab had CD19+ and CD20+ cell levels suppressed to zero (mm3) within one week. Recovery started for the subjects in the 100 mg placebo/active group after approximately 16 weeks (from these subjects' first infusion). In the 300 mg and 700 mg placebo/active groups, all subjects except one (700 mg) had persistent and complete CD19+ suppression at Week 48.

This study will evaluate the magnetic resonance imaging (MRI) efficacy and will investigate the safety of ofatumumab using a subcutaneous (SQ) formulation in subjects with RRMS. This Phase II study will be a multi-center, randomized, double-blind, placebo-controlled, dose ranging study in subjects with RRMS. Randomization will be stratified based on the absence or presence of GdE brain lesions present at screening. The core 54 week period of the study is made up of an up to 6-week Screening Phase, a 24-week Treatment Phase, and a 24-week Follow-up Phase. Subjects will attend the clinic a total of approximately twelve times (including Screening) during this core 54-week period of the study. Subjects who have remained enrolled and participate in the study from Screening though the end of the 24-Week Follow-Up Period (Week 48 Visit) will be considered completers. Upon completion or withdrawal from the core study period, subjects will be followed in the Individualized Follow-up Phase. Subjects will return to the clinic every 12 weeks for a B-cell count and other safety assessments. Subjects will remain in Individualized Follow-up (IFU) until CD19+ B-lymphocyte counts recover to LLN or baseline (if <LLN);OR if B-cell counts have not recovered by the Week 120 visit (100 weeks after the last possible treatment dose at Week 20), until either the B-cell counts or circulating IgG are >LLN or baseline levels (if <LLN). Male and female subjects with a diagnosis of RRMS will be screened for eligibility for the study. All non-MRI screening procedures should generally be completed within 14 days of informed consent being given. To the extent possible, investigators are to verify subjects meet all non MRI-related entry criteria before performing screening MRIs. Subjects who meet all inclusion and exclusion criteria will be centrally randomized into the study at the Baseline Visit (Week 0) to receive one of the following treatment arms: SQ administration of ofatumumab 3 mg, 30 mg, or 60 mg every 12 weeks, 60 mg every 4 weeks, or placebo. Half of the subjects randomized to the 30 mg group, or to either of the 60 mg groups, will receive a 3 mg conditioning dose at Week 0. Based on tolerability observed in other indications, the 3 mg conditioning dose may produce a more gradual lysis of B-cells, thereby reducing the cytokine release reactions to the initial 30 mg or 60 mg dose and potentially improve tolerability for subjects. The Treatment Phase lasts for 24 weeks and the subject will be seen 8 times during this phase. Upon completion or discontinuation of the Treatment Phase, subjects will enter a 24-week Follow-up Phase, during which they will not receive investigational product. Ideally, no other MS disease-modifying therapies should be taken during this period in order to allow for a clean analysis of safety data and the potential for Cluster of Differentiation (CD)+19 B-lymphocyte cell and immunoglobulin normalization to be assessed. However, if the start of a MS disease-modifying therapy is considered medically necessary, follow up will continue through the completion of the 24-Week Follow-up Phase. The subject will then be withdrawn from the study, and will not enter into the Individualized Follow-up Phase. Upon completion of the 24-Week Follow-up Phase, all subjects who have not started an MS disease modifying therapy (DMT) will enter the Individualized Follow up. During this Phase, subjects will return to the clinic every 12 weeks for a B-cell count and other safety assessments. If a subject starts a MS DMT during this follow-up phase they will be withdrawn from the study. To the extent possible, subjects experiencing a relapse during the study should return immediately to the clinic for evaluation. All MRI scans will be sent to a central reader for analysis. An Independent Data Monitoring Committee (IDMC) will evaluate risks relative to benefits through review of safety and efficacy information on an ongoing basis during the study. Approximately 245 subjects will be screened to provide around 196 subjects for randomization into the study. Assuming an attrition rate of 10% between the baseline visit and the six-month treatment visit, this will provide approximately 176 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed, written informed consent to participate in the study
* 18-55 years of age.
* Definite diagnosis of MS according to the 2010 revisions of the McDonald diagnostic criteria for MS [Polman, 2011].
* Subjects do not have any manifestation of another type of MS other than RRMS.
* Subjects must have a relapsing-remitting course of disease with at least one of the following prior to screening:
* At least one confirmed relapse within the previous year or
* At least two confirmed relapses within the previous 2 years or
* At least one relapse in the previous 2 years, with a GdE brain lesion on an MRI scan in the past year.
* Expanded Disability Status Scale (EDSS) score of 0-5.5 (inclusive) at screening.
* Neurologically stable with no evidence of relapse for at least 30 days prior to start of Screening and during the Screening Phase (subjects who relapse during the screening Phase can be re-screened, once the relapse has resolved).
* A female subject is eligible to enter the study if she is:
* Of non-childbearing potential
* Of childbearing potential and NOT pregnant or nursing, has a negative serum pregnancy test at screening, and agrees to one of the following:
* Complete abstinence from intercourse for the period from consent into the study until 6 months after the last dose of investigational product; or,
* Consistent and correct use of one of the following acceptable methods of birth control for the period from consent into the study until 6 months after the last dose of investigational product:

Oral contraceptives (either combined or progesterone only) Injectable progesterone Levonorgestrel implants Estrogenic vaginal ring Percutaneous contraceptive patches Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of <1% per year Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study; this male must be the sole partner for the subject Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).

A female is considered "Non-childbearing potential" if she is status-post hysterectomy, status-post surgical removal of both ovaries, has current, documented tubal ligation, or is postmenopausal and >2 years without menses. Female subjects who are post-menopausal <2 years must be confirmed menopausal by Follicle Stimulating Hormone (FSH) and estradiol levels.

A female is considered "childbearing potential" if she has functional ovaries, ducts, and uterus with no impairment that would cause sterility. This includes women with oligomenorrhea (even severe), and women who are perimenopausal or who have just begun to menstruate.

* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

* Unable to undergo MRI scans (e.g. due to pacemaker, severe claustrophobia, hypersensitivity to contrast media, or who lack adequate peripheral venous access).
* Any clinically significant brain abnormality other than MS found on MRI.
* Neurological findings consistent with Progressive Multifocal Leukoencephalopathy (PML) or confirmed PML (see Appendix 4, Section 11.4, for PML monitoring algorithm).
* Subjects whom experience a relapse during the Screening Phase. These subjects may be eligible for re-screening after consultation with GlaxoSmithKline (GSK).
* History of clinically significant Central Nervous System (CNS) trauma (e.g. traumatic brain injury, cerebral contusion, spinal cord compression) or a history or presence of myelopathy due to spinal cord compression by disk or vertebral disease.
* Prior treatment with any of the following:
* Systemic glucocorticoids or Adrenocorticotrophic hormone (ACTH) within one month prior to screening
* Receipt of a live vaccine within 6 weeks prior to screening
* Glatiramer acetate (Copaxone) or Interferon (IFN)-β (Betaferon, Betaseron, Avonex, or Rebif) within 3 months prior to screening
* Any immunomodulatory therapies, excluding glatiramer acetate or IFN-β, within 6 months prior to screening including natalizumab and fingolimod (Gilenya), immunoglobulin, or plasma exchange/plasmapheresis
* Any monoclonal antibodies at any time, other than natalizumab (Tysabri)
* Any lymphocyte-depleting therapies, including, but not limited to: cladribine, anti-Cluster of Differentiation 4 (CD4), total body irradiation, or bone marrow transplantation
* Any immunosuppressive agents, including, but not limited to: mitoxantrone, azathioprine, cyclosporine, cyclophosphamide, or tacrolimus
* Past or current history of medically significant adverse effects (including allergic reactions) from:
* Cetirizine (or equivalent)
* Paracetamol/acetaminophen
* Corticosteroids
* Known hypersensitivity to components of the investigational product.
* Past or current malignancy, except for
* Cervical carcinoma Stage 1B (cancer is present but has not spread) or less
* Non-invasive basal cell and squamous cell skin carcinoma
* Cancer diagnoses with a duration of complete response (remission) >5 years
* A history of hematologic malignancy excludes a subject from participation, regardless of response.
* Electrocardiogram (ECG) showing a clinically significant abnormality at Screening or showing an average QT interval for heart rate corrected using Bazett's Formula (QTcB) or QT interval for heart rate corrected using Fridericia's Formula (QTcF) interval >/=450 msec (>/=480 msec for subjects with a Bundle Branch Block) over 3 consecutive ECGs.
* Significant concurrent, uncontrolled medical condition including, but not limited to, cardiac, renal, hepatic, hematological, gastrointestinal, endocrine, immunodeficiency syndrome, pulmonary, cerebral, psychiatric, or neurological disease which in the opinion of the investigator could affect the subject's safety, impair the subject's reliable participation in the trial, impair the evaluation of endpoints, or necessitate the use of medication not allowed by this protocol.
* History of severe, clinically significant CNS trauma (e.g. cerebral contusion, spinal cord compression) or a history or presence of myelopathy due to spinal cord compression by disk or vertebral disease.
* Chronic or ongoing active infectious disease requiring long term systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, or active hepatitis C.
* Previous serious opportunistic or atypical infections.
* Positive polymerase chain reaction (PCR) screening for John Cunningham (JC) Virus as measured by plasma John Cunningham Virus (JCV) DNA.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
* Prior history, or suspicion, of tuberculosis (TB)
* Known history of positive serology for HIV.
* Any of the following screening laboratory values:
* White blood cells (WBC) <3.8 GI/L.
* Neutrophils <2 x 109/L.
* Platelets <1.3 x 105 GI/L.
* Circulating IgG, Immunoglobulin M (IgM), or Immunoglobulin A (IgA) levels < lower limit of normal (according to central laboratory range)
* Alanine aminotransferase (ALT) >2.0 times the upper limit of normal
* Aspartate aminotransferase (AST) >2.0 times the upper limit of normal
* Alkaline phosphatase (ALP) >1.5 times the upper limit of normal
* Bilirubin >1.5 times the upper limit of normal
* CD4 count <500 cells/mm3.
* CD19+ B-lymphocyte counts < lower limit of normal (according to central laboratory range)
* Creatinine clearance <60 mL/minute (by Cockcroft and Gault).
* Subjects known or suspected of not being able to comply with a trial protocol (e.g. due to alcoholism, drug dependency or psychological disorder).
* A documented history of attempted suicide over the 6 months prior to the screening visit, presents with suicidal ideation of type 4 or 5 on the C-Suicide Severity Rating Scale (SSRS) at the Screening visit, OR if in the investigator's judgment, the subject is at risk for a suicide attempt.
* Use of an investigational drug or other experimental therapy for a condition other than MS within 4 weeks, 5 pharmacokinetic half lives or duration of biological effect (whichever is longer) prior to screening. Any prior use of an investigational drug or other experimental therapy for MS at any time should be discussed with the GSK Medical Monitor.
* Current participation in any other interventional clinical trial. Participation in a non-interventional trial requires approval of the protocol by the GSK Medical Monitor
* French subjects: the French subject has participated in any study using an investigational drug during the previous 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 232 (Actual)
Dates: Start 2011-11-01; Primary Completion 2013-08-23 (Actual); Study Completion 2015-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (50):
- United States (16):
  - GSK Investigational Site, Cullman, Alabama
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Fairfield, Connecticut
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Sunrise, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Northbrook, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Round Rock, Texas
  - GSK Investigational Site, Seattle, Washington
- GSK Investigational Site, Sofia, Bulgaria
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Montreal, Quebec
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Jihlava
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Teplice
- GSK Investigational Site, Koebenhavn Ø, Denmark
- Germany (8):
  - GSK Investigational Site, Alzenau in Unterfranken, Bavaria
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (2):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Verona, Veneto
- Netherlands (2):
  - GSK Investigational Site, Sittard-geleen
  - GSK Investigational Site, Venray
- GSK Investigational Site, Hamar, Norway
- Russia (5):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
- Spain (8):
  - GSK Investigational Site, Baracaldo/Vizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Seville

REFERENCES:
- [Derived] Bar-Or A, Grove RA, Austin DJ, Tolson JM, VanMeter SA, Lewis EW, Derosier FJ, Lopez MC, Kavanagh ST, Miller AE, Sorensen PS. Subcutaneous ofatumumab in patients with relapsing-remitting multiple sclerosis: The MIRROR study. Neurology. 2018 May 15;90(20):e1805-e1814. doi: 10.1212/WNL.0000000000005516. Epub 2018 Apr 25. PMID 29695594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A participant (par.) completed the study if he/she completed all assessments up to and including the 24 Week Follow-up Phase (FUP) (Week 48) without prematurely discontinuing.
Pre-assignment Details: A total of 324 par. with Relapsing-Remitting Multiple Sclerosis (RRMS) were screened and 232 par. were randomized to 24 Week Treatment Phase (Weeks 0-12 were placebo controlled) of the study. A total of 231 par. received at least one dose of double-blind Investigational Product (IP) and were included in the Safety Population.
Groups:
- Placebo/Ofatumumab 3 mg: Par. received ofatumumab matching placebo subcutaneous (SC) injection every 4 weeks (q4w) from Week 0 to Week 20, except on Week 12 participants received 3 milligrams (mg) ofatumumab SC injection. Participants also received pre-medication of acetaminophen 1 gram (g) and antihistamine (cetirizine or equivalent) 10 mg prior to administration of each SC injection of investigational product.
- Ofatumumab 3 mg q12w: Par. received ofatumumab 3 mg SC injection every 12th week (q12w) on Week 1 and Week 12. Participants received matching placebo on Weeks 0, 4, 8, 16 and 20. Participants also received pre-medication of acetaminophen 1 g and antihistamine (cetirizine or equivalent) 10 mg prior to administration of each SC injection of investigational product.
- Ofatumumab 30 mg q12w: Par. received ofatumumab 3 mg conditioning dose SC injection or matching placebo on Week 0 and received ofatumumab 30 mg SC injection q12w on Week 1 and Week 12. Participants received matching placebo on Weeks 4, 8, 16 and 20. Participants also received pre-medication of acetaminophen 1 g and antihistamine (cetirizine or equivalent) 10 mg prior to administration of each SC injection of investigational product.
- Ofatumumab 60 mg q12w: Par. received ofatumumab 3 mg conditioning dose SC injection or matching placebo on Week 0 and received ofatumumab 60 mg SC injection q12w on Week 1 and Week 12. Participants received matching placebo on Weeks 4, 8, 16 and 20. Participants also received pre-medication of acetaminophen 1 g and antihistamine (cetirizine or equivalent) 10 mg prior to administration of each SC injection of investigational product.
- Ofatumumab 60mg q4w: Par. received ofatumumab 3 mg conditioning dose SC injection or matching placebo on Week 0 and received ofatumumab 60 mg SC injection q4w from Week 1 to Week 20. Participants also received pre-medication of acetaminophen 1 g and antihistamine (cetirizine or equivalent) 10 mg prior to administration of each SC injection of investigational product.
Period: Treatment Phase (Weeks 0-24)
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Started | 67 | 34 | 32 | 34 | 64
Completed to Week 12 | 65 | 31 | 30 | 33 | 60
Completed | 64 | 29 | 30 | 33 | 58
Not Completed | 3 | 5 | 2 | 1 | 6
Not completed — Adverse Event | 0 | 4 | 1 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1
Not completed — Other-Protocol defined stopping criteria | 1 | 1 | 0 | 0 | 2
Period: FUP (Weeks 24-48)
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Started (A total of 221 par. entered the FUP, including 7 of the 17 par. who were withdrawn before Week 24.) | 66 | 31 | 32 | 33 | 59
Completed | 63 | 30 | 30 | 32 | 57
Not Completed | 3 | 1 | 2 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 2
Period: Individualized FUP (Weeks 48+)
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Started (Par. whose CD19+ B lymphocyte counts had not recovered to lower limit of normal entered IFU phase.) | 16 | 18 | 16 | 20 | 42
Completed | 11 | 14 | 12 | 15 | 36
Not Completed | 5 | 4 | 4 | 5 | 6
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0
Not completed — Other-Protocol defined stopping criteria | 3 | 4 | 2 | 3 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Ofatumumab 3 mg: Par. received ofatumumab matching placebo SC injection q4w from Week 0 to Week 20, except on Week 12 participants received 3 mg ofatumumab SC injection. Participants also received pre-medication of acetaminophen 1 g and antihistamine (cetirizine or equivalent) 10 mg prior to administration of each SC injection of investigational product.
- Ofatumumab 3 mg q12w: Par. received ofatumumab 3 mg SC injection q12w on Week 1 and Week 12. Participants received matching placebo on Weeks 0, 4, 8, 16 and 20. Participants also received pre-medication of acetaminophen 1 g and antihistamine (cetirizine or equivalent) 10 mg prior to administration of each SC injection of investigational product.
- Total: Total of all reporting groups
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w | Total
Number analyzed (Participants) | 67 | 34 | 32 | 34 | 64 | 231
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (9.38) | 38.1 (8.29) | 37.2 (10.04) | 37.3 (9.67) | 36.2 (9.57) | 37.2 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 22 | 24 | 22 | 41 | 155
  Male | 21 | 12 | 8 | 12 | 23 | 76
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 0 | 0 | 0 | 1 | 2
  Asian - East Asian Heritage | 0 | 0 | 1 | 0 | 0 | 1
  White - White/Caucasian/European Heritage | 65 | 34 | 31 | 34 | 61 | 225
  Mixed Race | 1 | 0 | 0 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of New Gadolinium-enhancing (GdE) T1 Lesions at Week 12
Description: The cumulative number of new GdE T1 lesion at Week 12 were analyzed from screening based on magnetic resonance imaging (MRI) brain scans at Weeks 4, 8, and 12. The outcome measure was analyzed using an Emax model adjusting for the presence/absence of GdE lesions on the Screening MRI and assuming the number of new lesions followed a negative binomial distribution. Dose was fitted as a continuous variable. The number of scans contributing to the cumulative number of lesions was fitted as an offset. Estimates of the rate of cumulative number of new GdE lesions per scan at Week 12 were determined from the model. The all evaluable scans (AES) dataset was used which included all evaluable on-treatment MRI scans for each participant analysed.
Time Frame: Week 12
Population: Intent-to-Treat (ITT) Population comprised of all randomized par. who received at least one dose of IP and who had at least one post screen MRI assessment. Only those par. available at the specified time points were analyzed. Please see footnote of statistical analysis 1 for discrepancy in analysis population Week 24 and 48.
Measure: Mean (Standard Deviation); unit: Cumulative number of lesions
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 33 | 30 | 33 | 63
Cumulative number of lesions | 4.2 (7.57) | 1.7 (3.29) | 2.2 (3.41) | 2.2 (3.70) | 1.2 (2.83)
Statistical Analysis 1: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 3 mg q12w; Note: There is a discrepancy in the number of par. in ITT populations at Wk 24 and Wk 48: 228 and 229 respectively. This resulted from a data issue: one par was incorrectly excluded from ITT pop. at Wk 24, but correctly included in Wk 48. This error affects all source tables, analyses relating to ITT and per protocol populations, primary endpoint and secondary MRI endpoints reported at Wk 24. This discrepancy affects all statistical analyses, but not summary statistics; Test type: Superiority or Other; p < 0.001, Non-Linear Emax Model; Ratio = 0.35, 95% CI 2-sided [0.221 to 0.548]
Statistical Analysis 2: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 30 mg q12w; Test type: Superiority or Other; p < 0.001, Non-Linear Emax Model; Ratio = 0.35, 95% CI 2-sided [0.221 to 0.548]
Statistical Analysis 3: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60 mg q12w; Test type: Superiority or Other; p < 0.001, Non-Linear Emax Model; Ratio = 0.35, 95% CI 2-sided [0.221 to 0.548]
Statistical Analysis 4: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60mg q4w; Test type: Superiority or Other; p < 0.001, Non-Linear Emax Model; Ratio = 0.35, 95% CI 2-sided [0.221 to 0.548]

2. Secondary Outcome: Cumulative Number of New GdE T1 Lesions at Week 24
Description: The cumulative number of new GdE T1 lesion at Week 24 were analyzed from screen based on MRI brain scans at Weeks 4, 8, 12, 16, 20 and 24. Anticipating an underlying negative binomial distribution with a log-link function, adjusted for treatment and presence/absence of GdE lesions on the Screening MRI. Treatment group was fitted as a categorical variable. The number of scans contributing to the cumulative number of lesions was fitted as an offset. Estimates of the rate of cumulative number of new GdE T1 lesions per scan at Week 24 were determined from the model. The AES dataset was used which included all evaluable on-treatment MRI scans for each participant analyzed.
Time Frame: Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cumulative number of lesions
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 33 | 30 | 33 | 63
Cumulative number of lesions | 5.6 (9.34) | 2.2 (3.80) | 2.5 (3.88) | 2.2 (3.83) | 1.4 (3.04)
Statistical Analysis 1: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 3 mg q12w; Test type: Superiority or Other; p = 0.003, Generalized Linear Model; Ratio = 0.38, 95% CI 2-sided [0.20 to 0.72]
Statistical Analysis 2: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 30 mg q12w; Test type: Superiority or Other; p = 0.003, Generalized Linear Model; Ratio = 0.38, 95% CI 2-sided [0.20 to 0.72]
Statistical Analysis 3: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60 mg q12w; Test type: Superiority or Other; p = 0.001, Generalized Linear Model; Ratio = 0.35, 95% CI 2-sided [0.19 to 0.65]
Statistical Analysis 4: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60mg q4w; Test type: Superiority or Other; p < 0.001, Generalized Linear Model; Ratio = 0.23, 95% CI 2-sided [0.13 to 0.39]

3. Secondary Outcome: Change From Baseline in Brain Volume at Week 24 and Week 48
Description: Brain volume is a measure of brain size determined by a MRI scan. Baseline is defined as the par. last available assessment prior to initiation of the IP (i.e. Screening). Change from Baseline was calculated by subtracting the Baseline value from the post-Baseline value.
Time Frame: Baseline (Week 0), Week 24 and Week 48
Population: ITT Population. Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cubic centimeters
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 28 | 12 | 16 | 12 | 22
Cubic centimeters
  Week 24: number analyzed (Participants) | 25 | 12 | 16 | 12 | 22
  Week 24 | -13.5 (26.96) | -7.2 (22.26) | -8.4 (26.62) | -13.3 (34.02) | -1.4 (56.42)
  Week 48: number analyzed (Participants) | 28 | 12 | 16 | 11 | 19
  Week 48 | -22.0 (38.22) | -12.9 (14.55) | -5.0 (28.84) | -7.3 (29.16) | -11.8 (55.30)

4. Secondary Outcome: Cumulative Number of Persistent GdE Brain Lesions on T1-weighted MRI at Week 12
Description: The cumulative number of persistent GdE T1 lesions at Week 12 were analyzed from screen based on MRI scans at Weeks 4, 8, and 12. The AES dataset was used which included all evaluable on-treatment MRI scans for each par. analyzed.
Time Frame: Week 12
Population: ITT Population. Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Number of lesions per scan
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 34 | 30 | 33 | 63
Number of lesions per scan | 3.2 (7.41) | 1.2 (1.94) | 2.3 (3.94) | 1.8 (3.31) | 1.8 (4.81)

5. Secondary Outcome: Cumulative Number of All (New Plus Persistent) GdE Brain Lesions on T1-weighted MRI at Week 12
Description: The cumulative number of all (new plus persistent) GdE T1 lesion at Week 12 were analyzed from screen based on MRI brain scans at Weeks 4, 8 and 12. Anticipating an underlying negative binomial distribution with a log-link function, adjusted for treatment and presence/absence of GdE lesions on the Screening MRI. Treatment group was fitted as a categorical variable. The number of scans contributing to the cumulative number of lesions was fitted as an offset. Estimates of the rate of cumulative number of all (new plus persistent) GdE T1 lesions per scan at Week 12 were determined from the model. The AES dataset was used which included all evaluable on-treatment MRI scans for each par. analyzed.
Time Frame: Week 12
Population: ITT Population. Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cumulative number of lesions
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 33 | 30 | 33 | 63
Cumulative number of lesions | 7.4 (13.90) | 2.9 (4.62) | 4.5 (7.09) | 4.0 (6.70) | 3.1 (6.82)
Statistical Analysis 1: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 3 mg q12w; Test type: Superiority or Other; p < 0.001, Generalized Linear Model; Ratio = 0.31, 95% CI 2-sided [0.16 to 0.60]
Statistical Analysis 2: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 30 mg q12w; Test type: Superiority or Other; p = 0.075, Generalized Linear Model; Ratio = 0.56, 95% CI 2-sided [0.29 to 1.06]
Statistical Analysis 3: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60 mg q12w; Test type: Superiority or Other; p = 0.035, Generalized Linear Model; Ratio = 0.51, 95% CI 2-sided [0.27 to 0.95]
Statistical Analysis 4: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60mg q4w; Test type: Superiority or Other; p < 0.001, Generalized Linear Model; Ratio = 0.32, 95% CI 2-sided [0.19 to 0.55]

6. Secondary Outcome: Total Volume of New GdE Brain Lesions on T1-weighted MRI at Week 12
Description: Lesion volume is a measure of lesion size determined by a MRI brain scan. The cumulative volume of new GdE T1 lesions at Week 12 were analyzed from screen based on MRI brain scans at Weeks 4, 8 and 12. Anticipating an underlying negative binomial distribution with a log-link function, adjusted for treatment and presence/absence of GdE lesions on the Screening MRI. Treatment group was fitted as a categorical variable. The number of scans contributing to the cumulative volume of lesions was fitted as an offset. Estimates of the rate of cumulative volume of new GdE T1 lesions per scan at Week 12 were determined from the model. The AES dataset was used which included all evaluable on-treatment MRI scans for each par. analyzed.
Time Frame: Week 12
Population: ITT Population. Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cubic millimeter (mm^3)
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 34 | 30 | 33 | 63
Cubic millimeter (mm^3) | 607.5 (1090.89) | 226.5 (449.37) | 452.9 (682.33) | 248.6 (457.62) | 146.6 (304.89)
Statistical Analysis 1: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 3 mg q12w; Test type: Superiority or Other; p = 0.026, Generalized Linear Model; Ratio = 0.22, 95% CI 2-sided [0.06 to 0.84]
Statistical Analysis 2: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 30 mg q12w; Test type: Superiority or Other; p = 0.296, Generalized Linear Model; Ratio = 0.49, 95% CI 2-sided [0.13 to 1.86]
Statistical Analysis 3: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60 mg q12w; Test type: Superiority or Other; p = 0.285, Generalized Linear Model; Ratio = 0.50, 95% CI 2-sided [0.14 to 1.78]
Statistical Analysis 4: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60mg q4w; Test type: Superiority or Other; p = 0.009, Non-Linear Emax Model; Ratio = 0.25, 95% CI 2-sided [0.09 to 0.71]

7. Secondary Outcome: Total Volume of All (New and Persistent) GdE Brain Lesions on T1-weighted MRI at Week 12
Description: Lesion volume is a measure of lesion size determined by a MRI brain scan. The cumulative volume of all (new and persistent) GdE T1 lesions at Week 12 were analyzed from screen based on MRI brain scans at Weeks 4, 8 and 12. The endpoint was analyzed using a generalized linear model assuming an underlying negative binomial distribution with a log-link function, adjusted for treatment and presence/absence of GdE lesions on the Screening MRI. Treatment group was fitted as a categorical variable. The number of scans contributing to the cumulative volume of lesions was fitted as an offset. Estimates of the rate of cumulative volume of all (new and persistent) GdE T1 lesions per scan at Week 12 were determined from the model. The AES dataset was used which included all evaluable on-treatment MRI scans for each par. analyzed.
Time Frame: Week 12
Population: ITT Population. Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 33 | 30 | 33 | 63
mm^3 | 1039.6 (1809.97) | 386.2 (628.41) | 886.2 (1637.47) | 426.5 (679.44) | 344.4 (735.57)
Statistical Analysis 1: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 3 mg q12w; Test type: Superiority or Other; p = 0.004, Generalized Linear Model; Ratio = 0.18, 95% CI 2-sided [0.05 to 0.58]
Statistical Analysis 2: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 30 mg q12w; Test type: Superiority or Other; p = 0.248, Generalized Linear Model; Ratio = 0.50, 95% CI 2-sided [0.15 to 1.63]
Statistical Analysis 3: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60 mg q12w; Test type: Superiority or Other; p = 0.181, Generalized Linear Model; Ratio = 0.46, 95% CI 2-sided [0.15 to 1.43]
Statistical Analysis 4: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60mg q4w; Test type: Superiority or Other; p = 0.003, Generalized Linear Model; Ratio = 0.24, 95% CI 2-sided [0.10 to 0.62]

8. Secondary Outcome: Cumulative Number of New and Newly Enlarging GdE T2 Lesions at Week 12
Description: The cumulative number of new and newly enlarging GdE T2 lesions (NET2L) at Week 12 were analyzed from screen based on MRI brain scans at Weeks 4, 8 and 12. The endpoint was analyzed using a generalized linear model assuming an underlying negative binomial distribution with a log-link function, adjusted for treatment and presence/absence of GdE lesions on the Screening MRI. Treatment group was fitted as a categorical variable. The number of scans contributing to the cumulative number of lesions was fitted as an offset. Estimates of the rate of cumulative number of NET2L per scan at Week 12 were determined from the model. The AES dataset was used which included all evaluable on-treatment MRI scans for each par. analyzed.
Time Frame: Week 12
Population: ITT Population. Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cumulative number of lesions
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 33 | 30 | 33 | 63
Cumulative number of lesions | 3.7 (6.72) | 1.2 (2.38) | 1.6 (2.79) | 1.7 (2.67) | 0.8 (1.55)
Statistical Analysis 1: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 3 mg q12w; Test type: Superiority or Other; p < 0.001, Generalized Linear Model; Ratio = 0.29, 95% CI 2-sided [0.15 to 0.58]
Statistical Analysis 2: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 30 mg q12w; Test type: Superiority or Other; p = 0.002, Generalized Linear Model; Ratio = 0.34, 95% CI 2-sided [0.17 to 0.68]
Statistical Analysis 3: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60 mg q12w; Test type: Superiority or Other; p = 0.006, Generalized Linear Model; Ratio = 0.40, 95% CI 2-sided [0.21 to 0.77]
Statistical Analysis 4: Comparison: Placebo/Ofatumumab 3 mg vs Ofatumumab 60mg q4w; Test type: Superiority or Other; p < 0.001, Generalized Linear Model; Ratio = 0.19, 95% CI 2-sided [0.11 to 0.35]

9. Secondary Outcome: Total Volume of New and/or Newly Enlarging T2 Lesions at Week 12
Description: Lesion volume is a measure of lesion size determined by a MRI brain scan. T2 lesions, are indicative of brain myelin content.The cumulative volume of new and/or newly enlarging T2 lesions at Week 12 were analyzed from screen based on MRI brain scans at Weeks 4, 8, and 12. The AES dataset was used which included all evaluable on-treatment MRI scans for each par.
Time Frame: Week 12
Population: ITT Population. Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 34 | 30 | 33 | 63
mm^3 | 1204.5 (3426.79) | 279.9 (695.75) | 611.3 (1042.06) | 293.8 (576.35) | 167.9 (450.65)

10. Secondary Outcome: Cumulative Number of New T1 Hypointense Lesions at Week 24 and Week 48
Description: The cumulative number of new T1 hypointense lesions at week 24 were analyzed from screen based on MRI brain scans at Weeks 4, 8, 12, 16, 20 and 24. The AES dataset was used which included all evaluable on-treatment MRI scans for each par.
Time Frame: Week 24 and Week 48
Population: ITT Population. Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Number of lesions
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 34 | 32 | 33 | 63
Number of lesions
  Week 24: number analyzed (Participants) | 67 | 34 | 30 | 33 | 63
  Week 24 | 0.4 (0.96) | 0.4 (1.26) | 0.5 (1.01) | 0.5 (1.12) | 0.3 (0.78)
  Week 48 | 0.6 (1.27) | 0.5 (1.26) | 0.5 (0.98) | 0.6 (1.25) | 0.3 (0.96)

11. Secondary Outcome: Cumulative Volume of New T1 Hypointense Lesions at Week 24 and Week 48
Description: Lesion volume is a measure of lesion size determined by a MRI brain scan. Baseline is defined as the participant's last available assessment prior to initiation of IP. Change from Baseline was calculated by subtracting the Baseline value from the post-Baseline value. The AES dataset was used which included all evaluable on-treatment MRI scans for each par.
Time Frame: Baseline, Week 24 and Week 48
Population: ITT Population. Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
Number analyzed (Participants) | 67 | 34 | 32 | 33 | 63
mm^3
  Week 24: number analyzed (Participants) | 67 | 34 | 30 | 33 | 63
  Week 24 | 86.9 (240.40) | 43.1 (131.96) | 67.4 (147.00) | 65.0 (139.14) | 42.9 (140.93)
  Week 48 | 113.6 (270.89) | 54.2 (137.74) | 63.2 (143.14) | 116.3 (370.35) | 53.2 (173.62)

ADVERSE EVENTS:
Time Frame: On treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of administration of the study drug until the follow-up contact (up to Week 24).
Description: SAEs and non-serious AEs were reported for members of the safety population, comprised of all par. who were randomized to treatment, and received at least one dose of study medication.
Arm/Group | Placebo/Ofatumumab 3 mg | Ofatumumab 3 mg q12w | Ofatumumab 30 mg q12w | Ofatumumab 60 mg q12w | Ofatumumab 60mg q4w
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/34 | 0/32 | 0/34 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/34 | 0/32 | 1/34 | 4/64
Other Adverse Events (participants affected / at risk) | 41/67 | 20/34 | 23/32 | 22/34 | 47/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Ofatumumab 3 mg (N=67) | Ofatumumab 3 mg q12w (N=34) | Ofatumumab 30 mg q12w (N=32) | Ofatumumab 60 mg q12w (N=34) | Ofatumumab 60mg q4w (N=64)
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Ofatumumab 3 mg (N=67) | Ofatumumab 3 mg q12w (N=34) | Ofatumumab 30 mg q12w (N=32) | Ofatumumab 60 mg q12w (N=34) | Ofatumumab 60mg q4w (N=64)
Injection related reaction (Injury, poisoning and procedural complications) | 18 | 16 | 13 | 17 | 42
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 8 | 1 | 4 | 7 | 7
Urinary tract infection (Infections and infestations) | 4 | 3 | 3 | 2 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 7 | 2 | 2 | 2 | 6
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 4
Neuralgia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 8 | 0 | 3 | 2 | 3
Pyrexia (General disorders) | 2 | 2 | 2 | 1 | 1
Injection site pain (General disorders) | 0 | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0
Reticulocyte count decreased (Investigations) | 1 | 0 | 2 | 1 | 1
Blood immunoglobulin G decreased (Investigations) | 0 | 2 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The incorrect exclusion of one par. from ITT pop. at Wk 24 was not considered to impact overall interpretation of data: no updates were made to source tables/analyses. This par. had withdrawn early, having never received a dose of active study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.